CLINICAL TRIAL: NCT01181908
Title: A Study to Investigate the Psychomotor and Cognitive Effects of Alcohol When Co-administered With GSK1144814 or Matching Placebo in Healthy Subjects.
Brief Title: Alcohol Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 113476
Record Dates: First submitted 2009-12-17; First posted 2010-08-13 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Alcoholism
Keywords: alcohol; drug interaction; pharmacodynamic
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK1144814 (Experimental): Subjects will receive either GSK1144814 or placebo at each treatment arm.
  Interventions: Drug: single dose
- placebo (Placebo Comparator): Subjects will receive either GSK1144814 or placebo at each treatment arm.
  Interventions: Drug: single dose

INTERVENTIONS:
Drug: single dose — Subjects will receive a single dose of GSK1144814 or placebo.

SUMMARY:
The purpose of this study is understand the effects of GSK114814 and alcohol in healthy volunteers when taken together.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the CNS effects of co-administration of GSK1144814 with alcohol. Healthy volunteers who meet the eligibility criteria will be randomized to receive GSK1144814 or placebo with alcohol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female
* Body weight 50 kg or higher and BMI within the range 19 - 29.9 kg/m2
* Willing to use appropriate contraception methods

Exclusion Criteria:

* Positive HIV, Hepatitis B surface antigen or Hepatitis C antibody result
* Any serious medical disorder or condition
* Any history of an endocrine disorder.
* Any clinically significant laboratory abnormality.
* History of psychiatric illness.
* Any history of suicidal attempts or behavior.
* Positive urine drug screen or positive blood alcohol
* Pregnant, nursing or potential to have a child
* Past history of alcohol dependence or abuse.
* History of increased sensitivity to the effects of alcohol or violent behaviour/aggression when intoxicated.
* smokers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-11-11 (Actual); Primary Completion 2009-12-30 (Actual); Study Completion 2009-12-30 (Actual)

PRIMARY OUTCOMES:
pharmacodynamic measures for various psychomotor/cognition function and subjective effects | pre and post study drug administration

SECONDARY OUTCOMES:
alcohol level | during and post alcohol administration
blood level of GSK1144814 | pre and post study drug administration
safety and tolerability as measured by adverse events, vital signs, clinical laboratory measurements and validated clinical assessment scales | throughout the study pre- and post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Leiden, Netherlands

REFERENCES:
- [Background] te Beek ET, Hay JL, Bullman JN, Burgess C, Nahon KJ, Klaassen ES, Gray FA, van Gerven JM. Pharmacokinetics and central nervous system effects of the novel dual NK1 /NK3 receptor antagonist GSK1144814 in alcohol-intoxicated volunteers. Br J Clin Pharmacol. 2013 May;75(5):1328-39. doi: 10.1111/bcp.12004. PMID 23067311
- See also: Results for study 113476 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113476?search=study&study_ids=113476#rs